CLINICAL TRIAL: NCT06720181
Title: Functional Evaluation of Brain Pain Centers in Endometriosis-Associated Chronic Pelvic Pain Exploring the Impact of Central Sensitization Using a Novel MRI Technique: A Retrospective Study
Brief Title: Functional Evaluation of Brain Pain Centers in Endometriosis-Associated Chronic Pelvic Pain Exploring the Impact of Central Sensitization Using a Novel MRI Technique
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Isin ERDOGAN, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IE1
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Novel MRI Technique
Keywords: chronic pelvic pain; endometriosis; brain pain centers; functional connectivity
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with chronic pelvic pain and deep infiltrating endometriosis
  Interventions: Diagnostic Test: MRI
- Group 2: Patients with cystic endometriosis (ovarian endometriomas) without chronic pelvic pain
  Interventions: Diagnostic Test: MRI
- Group 3: Women with no gynecological pathology, under routine outpatient follow-up, matched for age and body mass index
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Resting-state Functional Magnetic Resonance Imaging and Diffusion Tensor Magnetic Resonance Imaging of the brain

SUMMARY:
Endometriosis is a chronic inflammatory disease characterized by the presence of endometrial tissue outside the uterus, affecting about 10% of reproductive-age women. It is commonly associated with chronic pelvic pain, present in 40-50% of women with persistent pelvic pain and 30-40% of infertile women. The condition contributes to chronic pain through mechanisms like inflammation, neurogenic inflammation, neuroangiogenesis, and central sensitization.

Central sensitization involves changes in brain function and can be assessed using magnetic resonance imaging (MRI). While studies have shown the role of brain changes in chronic pain for conditions like migraine and fibromyalgia, research on pain chronicization in endometriosis is limited.

This study focuses on evaluating functional changes in brain pain centers associated with endometriosis-related chronic pelvic pain using neuroimaging. The goal is to enhance understanding of the pathophysiology of chronic pain and emphasize the potential of MRI in guiding more effective management strategies for endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic disease defined by the presence of endometrial stroma and glands outside the uterus. It affects approximately 10% of women of reproductive age and is detected in 40-50% of women experiencing persistent pelvic pain and 30-40% of infertile women. Clinically classified as an inflammatory and systemic disease, endometriosis often manifests as pelvic pain. It is believed that endometriosis contributes to chronic pelvic pain through mechanisms such as inflammation, neurogenic inflammation, neuroangiogenesis, peripheral sensitization, central sensitization, and cross-organ sensitization.

Central sensitization can be identified by evaluating functional changes in the brain using magnetic resonance imaging (MRI). Numerous studies have demonstrated the importance of brain functional changes in the chronicization of pain in various conditions, including migraine, fibromyalgia, trigeminal neuralgia, and chronic lower back pain. However, there are limited MRI studies investigating the chronicization of pain associated with endometriosis.

In this study, we aim to highlight the benefits of neuroimaging in elucidating the pathophysiology of chronic pain by examining the functional changes in brain pain centers in chronic pelvic pain associated with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18-45 who underwent brain magnetic resonance imaging, including those with endometriosis and those without gynecological pathology, matched for age and body mass index

Exclusion Criteria:

patients who were pregnant patients in the postmenopausal period patients who had detected pathologies in brain imaging

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The medical records of patients who visited the Gynecology Outpatient Clinic and/or were hospitalized in the Gynecology Department of Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, between June 1, 2022, and September 1, 2023, were reviewed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Neuroimaging in patients suffered from endometriosis-associated chronic pelvic pain | baseline
  The functional connectivity of brain regions involved in pain pathophysiology, including the anterior and posterior segments of the anterior cingulate gyrus, insula, thalamus, and amygdala, with other brain areas was investigated using the seed-to-voxel connectivity method.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No